CLINICAL TRIAL: NCT07259057
Title: Effects of Erector Spinae Plane Block on Postoperative Systemic Functions in Patients Undergoing Open-Heart Surgery Via Sternotomy
Brief Title: Erector Spinae Plane Block and Postoperative Recovery After Open-Heart Surgery
Acronym: ESPB-SYSHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, Assistant Professor, Department of Anesthesiology and Critical Care, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KTU-ESPB-2022-247
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain Management; Open-heart Surgery; Median Sternotomy; Erector Spinae Plane Block
Keywords: Erector Spinae Plane Block; Regional Anesthesia; Open-Heart Surgery; Postoperative Pain; Postoperative Recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group randomized controlled design in which participants were allocated in a 1:1 ratio to receive either bilateral erector spinae plane block (ESPB) before anesthesia induction or standard intravenous opioid-based analgesia. Both groups were followed concurrently throughout the perioperative and postoperative periods for outcome assessment.
Masking Description: This study was conducted as an open-label randomized controlled trial. Neither participants nor care providers nor investigators were blinded to group allocation because the erector spinae plane block procedure is a hands-on regional anesthesia technique that cannot be feasibly masked. Outcome assessors were also not blinded due to the nature of the intervention and perioperative workflow.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (ESPB) (Experimental): Patients received bilateral ultrasound-guided erector spinae plane block at the T5 level before induction of general anesthesia. A total of 20 mL of 0.25% bupivacaine was injected on each side.
  Interventions: Procedure: Erector spinae plane block (ESPB)
- Intravenous Opioid Analgesia (Control) (Active Comparator): Standard intravenous opioid-based analgesia administered without regional block.
  A fentanyl infusion (0.5 μg/kg/h) was initiated immediately after induction of general anesthesia and continued intraoperatively per institutional protocol.
  Interventions: Drug: Intravenous Opioid Analgesia

INTERVENTIONS:
Procedure: Erector spinae plane block (ESPB) — Bilateral ultrasound-guided erector spinae plane block performed at the T5 vertebral level before induction of general anesthesia.
  A total of 20 mL of 0.25% bupivacaine was injected between the erector spinae muscle and the transverse process on each side using a high-frequency linear ultrasound probe and a 22-gauge needle.
  Arms: Erector Spinae Plane Block (ESPB)
Drug: Intravenous Opioid Analgesia — Standard intravenous opioid-based analgesia administered without regional block. Fentanyl infusion (0.5 μg/kg/h) was started after induction and continued intraoperatively according to institutional protocol.
  Arms: Intravenous Opioid Analgesia (Control)

SUMMARY:
This prospective randomized controlled clinical trial evaluated the effects of bilateral erector spinae plane block (ESPB) on postoperative systemic functions in adult patients undergoing elective open-heart surgery via median sternotomy. Sixty-six participants were randomized to receive either bilateral ultrasound-guided ESPB before anesthesia induction or standard intravenous opioid analgesia. Postoperative outcomes-including pain scores, rescue analgesic requirements, hemodynamic parameters, respiratory variables, and laboratory values-were monitored for forty-eight hours. The study was conducted to determine whether ESPB provides improved postoperative pain control and supports systemic recovery compared with intravenous opioid-based analgesia.

DETAILED DESCRIPTION:
Open-heart surgery performed through median sternotomy is associated with significant postoperative pain, sympathetic activation, respiratory impairment, and delayed recovery. Conventional postoperative analgesia, primarily based on intravenous opioids, may provide adequate pain relief but is frequently limited by adverse effects such as sedation, nausea, respiratory depression, and hemodynamic fluctuations. Therefore, safer and more effective multimodal analgesia strategies are required for cardiac surgical patients.

The erector spinae plane block (ESPB) is a paraspinal interfascial block that allows the spread of local anesthetic to the dorsal and ventral rami, intercostal nerves, and paravertebral region, providing both somatic and visceral analgesia. ESPB has been increasingly used as an alternative to thoracic epidural analgesia, especially in patients undergoing cardiac surgery where neuraxial techniques may pose risks related to anticoagulation and sympathetic blockade.

This prospective randomized controlled clinical trial was designed to evaluate whether bilateral ultrasound-guided ESPB can improve postoperative systemic functions in patients undergoing elective open-heart surgery via sternotomy. A total of sixty-six adults classified as ASA II-III were randomized into two groups. The intervention group received bilateral ESPB at the T5 level using twenty milliliters of 0.25% bupivacaine per side prior to induction of general anesthesia, whereas the control group received standard intravenous opioid-based analgesia.

Postoperative outcomes were monitored for forty-eight hours and included pain scores measured by the Numeric Rating Scale (NRS), time to rescue analgesia, total analgesic consumption, hemodynamic parameters, respiratory measurements, and laboratory markers such as hemoglobin, creatinine, AST, and ALT. The primary objective was to determine whether ESPB provides superior postoperative pain control compared with intravenous opioid analgesia. Secondary objectives included assessing the effects of ESPB on hemodynamic stability, respiratory recovery, and systemic laboratory parameters.

The study was conducted after ethics committee approval, and written informed consent was obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* Scheduled for elective open-heart surgery via median sternotomy (CABG or valve surgery)
* ASA physical status II-III
* Provided written informed consent
* BMI < 35 kg/m²

Exclusion Criteria:

* Age <18 or >75 years
* Known coagulopathy or anticoagulation contraindicating regional block
* Infection or dermatological lesion at the injection site
* Allergy to local anesthetics
* Chronic use of opioids, anticonvulsants, antidepressants, or corticosteroids
* Significant psychiatric or cognitive disorder preventing cooperation
* Severe arrhythmia or hemodynamic instability prior to surgery
* Local anesthetic toxicity risk factors or anatomic deformity preventing block placement
* Non-elective or emergency cardiac surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (NRS Score) | First 12 hours after extubation (measured at 1, 6, and 12 hours)
  Pain intensity will be assessed using the Numeric Rating Scale (NRS; 0 = no pain, 10 = worst imaginable pain) at standardized postoperative time points.

SECONDARY OUTCOMES:
Time to First Rescue Analgesic Requirement | Within 48 hours post-extubation
  Time in hours from extubation to first administration of rescue analgesia (tramadol or diclofenac).
Total Rescue Analgesic Consumption | 48 hours post-extrubation
  Total amount of rescue analgesics administered (mg of tramadol and diclofenac) during the first 48 postoperative hours.
Heart Rate (beats per minute) | First 24 postoperative hours
  Heart rate (HR) values recorded at predefined postoperative intervals.
Mobilization Time | Up to postoperative day 3
  Time from ICU admission to first successful mobilization (sitting or standing with assistance).
Length of Hospital Stay | From completion of surgery until hospital discharge, up to 14 days.
  Total duration of postoperative hospitalization, measured in days.
Postoperative Hemoglobin Change | 24 hours after surgery
  Difference between preoperative and postoperative hemoglobin levels (g/dL).
Serum Creatinine Level (mg/dL) | Preoperative baseline and postoperative 24 hours (up to 24 hours after surgery).
  Serum creatinine concentration will be measured as an indicator of postoperative renal function. Values are reported in milligrams per deciliter (mg/dL). Higher values indicate worse renal function.
Mean Arterial Pressure (mmHg) | First 24 postoperative hours
  Mean arterial pressure (MAP) values recorded at predefined postoperative intervals.
Urine Output (mL/kg/hour) | First 24 hours after surgery (up to 24 hours postoperative).
  Urine output will be measured as an indicator of renal perfusion and early postoperative renal function. Values are reported in milliliters per kilogram per hour (mL/kg/h). Higher values indicate better renal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Farabi Hospital, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarica F, Erturk E, Kutanis D, Akdogan A, Senel AC. Comparison of Thoracic Epidural Analgesia and Traditional Intravenous Analgesia With Respect to Postoperative Respiratory Effects in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 Jun;35(6):1800-1805. doi: 10.1053/j.jvca.2020.09.110. Epub 2020 Sep 20. PMID 33059978
- [Result] Oostvogels L, Weibel S, Meissner M, Kranke P, Meyer-Friessem CH, Pogatzki-Zahn E, Schnabel A. Erector spinae plane block for postoperative pain. Cochrane Database Syst Rev. 2024 Feb 12;2(2):CD013763. doi: 10.1002/14651858.CD013763.pub3. PMID 38345071
- [Result] Shan XS, Liao DW, Guo J, Xia ZY, Lv X, Shen J, Tong JH, Wei FJ, Li XS, Qu XF, Wang XB, Wang YB, Ou SS, Yang YF, Meng L, Liu H, Peng K, Ji FH. Effect of liposomal bupivacaine for preoperative erector spinae plane block on postoperative pain following video-assisted thoracoscopic lung resection: a multicenter, randomized, double-blind, clinical trial. Int J Surg. 2025 Nov 11. doi: 10.1097/JS9.0000000000003956. Online ahead of print. PMID 41217370